CLINICAL TRIAL: NCT02312219
Title: Imaging Companion Study To ACTG A5314: Effect of Reducing Inflammation With Low Dose Methotrexate on Inflammatory Markers and Endothelial Function in Treated and Suppressed HIV Infection
Brief Title: PET/CT Imaging Companion Study To ACTG A5314
Acronym: PET/CTMTX
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Harvard School of Public Health (HSPH) (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ahmed Tawakol, Director: Integrative BioImaging Trials, Massachusetts General Hospital
Other Study IDs: 2014P000145
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2018-09

CONDITIONS: HIV; Inflammation; Atherosclerosis
Keywords: HIV; Inflammation; Atherosclerosis; Positron-Emission Tomography; Imaging; fluorodeoxyglucose
MeSH Terms: conditions — Inflammation; Atherosclerosis | interventions — Folic Acid; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low Dose Methotrexate: Subjects will take 1 mg folic acid once daily plus 5 mg methotrexate (MTX) . If clinically stable at the week 1 visit, the dose of MTX will be increased to 10 mg once weekly through week 12. For subjects who remain clinically stable on 10 mg MTX or placebo through the week 12 visit, the dose of MTX will be increased to 15 mg once weekly through week 24. If the subject does not meet the criteria for dose escalation at the week 1 or 12 study visit, then the subject will remain on his/her current dose until the next study visit at which time he/she will be re-evaluated for dose escalation.
  Interventions: Drug: Folic Acid; Drug: Low Dose Methotrexate
- Placebo: Subjects will take 1 mg folic acid once daily plus placebo once weekly. If clinically stable at weeks 1 and 12, the number of placebo tablets will be increased in a manner matching those on the MTX.
  Interventions: Drug: Folic Acid; Drug: Placebo

INTERVENTIONS:
Drug: Folic Acid — 1 mg folic acid once daily
  Other Names: Folate
Drug: Placebo — placebo once weekly
  Other Names: (Placebo for MTX)
  Groups: Placebo
Drug: Low Dose Methotrexate — An anti-inflammatory drug
  Other Names: Methotrexate
  Groups: Low Dose Methotrexate

SUMMARY:
HIV-infected individuals on antiretroviral therapy (ART) are at increased risk for cardiovascular disease (CVD), likely due to chronically increased inflammation. Low-dose methotrexate (LDMTX) may reduce CVD risk in people with rheumatoid arthritis, who like those with HIV, have increased levels of inflammation. The NHLBI is funding a clinical trial targeting the excess inflammation in HIV. That "Parent Study" is a randomized, double-blind, placebo-controlled trial (NCT01949116) that will assess whether 24-week treatment with LDMTX: i) is safe, ii) reduces circulating inflammatory biomarkers and levels of immune cell activation and iii) improves brachial artery reactivity. However, neither the biomarkers nor endothelial function tests measured as part of the parent study will report on atherosclerotic inflammation, (the desired pathobiological target of LDMTX therapy in HIV). As such, the direct evaluation of arterial inflammation would substantially enhance the scientific value of the trial. In this imaging sub-study, the overall goal is to determine if treating virologically suppressed, HIV-infected individuals with LDMTX will reduce inflammation within the arterial wall.

This fully integrated ancillary study would, in a subset of patients enrolled in the parent trial: (i) assess the impact of LDMTX on arterial inflammation, (ii) evaluate mechanisms responsible for arterial inflammation in HIV and iii) explore mechanisms responsible for actions of LDMTX on the artery wall. Accordingly, the proposed study would provide unique and highly complementary information that would greatly increase the knowledge and mechanistic insights gained from Parent Study. The ancillary study has two specific aims1) To determine the impact of anti-inflammatory treatment with LDMTX on arterial inflammation, as assessed by FDG-PET/CT imaging, in virally suppressed HIV-infected individuals., and 2) To evaluate the cellular and biochemical basis of the effect of LDMTX therapy on arterial inflammation in HIV.

DETAILED DESCRIPTION:
HIV infection is associated with a substantially increased risk of CVD that is not fully accounted for by traditional risk factors. Several lines of evidence suggest that chronic immune cell activation may be complicit. In support of this concept, we recently used 18F-FDG-PET/CT to demonstrate that HIV-infected individuals have increased arterial inflammation compared to non-HIV, FRS-matched controls and that the degree of arterial inflammation is related to markers of monocyte activation. Further, we and others have shown that increased arterial FDG uptake predicts future CVD events in non-HIV cohorts. Together, these observations support the concept that targeting arterial inflammation may provide benefit for HIV infected individuals.

The NHLBI recently provided funding for a clinical trial targeting the excess inflammation in HIV. The "Parent Study" is being performed as a collaboration with the National Institute of Allergy and Infectious Diseases (NIAID) AIDS Clinical Trials Group and the NHLBI. That randomized, double-blind, placebo-controlled trial will assess whether 24-week treatment with very low-dose methotrexate (LDMTX): i) is safe, ii) reduces levels of circulating inflammatory biomarkers and activated immune cells and iii) improves brachial artery reactivity (BART). However, neither the biomarkers nor the BART studies measured as part of Parent Study will report on atherosclerotic inflammation, (the desired pathobiological target of LDMTX therapy in HIV). As such, the direct evaluation of arterial inflammation would substantially enhance the scientific value of the Parent Study.

Atherosclerotic inflammation can be non-invasively and reproducibly measured with FDG-PET/CT imaging, a well-validated quantitative technique that can sensitively detect changes in atherosclerotic inflammation. FDG-PET/CT imaging has been employed in several multi-center trials to measure changes in arterial inflammation in response to anti-inflammatory treatments. Accordingly, we propose a time sensitive ancillary imaging study to determine if treating virologically suppressed, HIV-infected individuals with LDMTX reduces atherosclerotic inflammation, assessed by FDG-PET/CT. Our central hypothesis is that persistent immune cell activation results in chronic arterial inflammation, which subsequently contributes to the CVD risk observed in HIV. This fully integrated ancillary study would, in a subset of patients enrolled in the parent trial: (i) assess the impact of LDMTX on arterial inflammation, and (ii) identify the immune cell subtypes whose changes (with LDMTX) are associated with changes in arterial inflammation. Accordingly, the proposed ancillary study would provide unique and highly complementary information that would greatly increase the knowledge and mechanistic insights gained from the Parent Study. The ancillary study has two specific aims:

Specific Aim 1: To determine the impact of anti-inflammatory treatment with LDMTX on arterial inflammation, as assessed by FDG-PET/CT imaging, in virally suppressed HIV-infected individuals. [Primary and secondary outcomes]

Knowledge Gap/Need: The parent study does not provide for assessment of the target pathology (arterial inflammation) hence insights regarding effects of LDMTX treatment on arterial inflammation are needed.

Hypothesis 1: LDMTX therapy will reduce arterial inflammation (to a greater extent than placebo).

To test hypothesis 1: We will determine in 91 patients (a subset of the parent study) if arterial inflammation (measured with PET/CT at 0 and 24 weeks) is reduced by LDMTX (relative to placebo).

Specific Aim 2: To evaluate the cellular and biochemical mediators associated with arterial inflammation in HIV and to explore the potential mechanism of the effect of LDMTX therapy on arterial inflammation in HIV. [Exploratory outcomes]

Knowledge Gap/Need: The parent study, on its own, does not provide the tools to directly evaluate arterial inflammation in HIV. Evaluation of the relationships between circulating inflammatory mediators and arterial inflammation in the context of this study would yeild mechanistic insights regarding atherosclerotic disease in HIV and provide a greater understanding of the effect of LDMTX on arterial inflammation in HIV.

Hypothesis 2.1:At baseline, arterial inflammation is closely associated with measures of activated immune cells (CD14+/CD16+ monocytes). Additional relationships might be seen between arterial inflammation and other cellular subsets (e.g. T-cells), inflammatory cytokines, and endothelial function.

Hypothesis 2.2: Post-treatment changes in arterial inflammation are positively correlated with changes in measures of activated immune cells (especially activated monocytes).

To test these hypotheses: We will evaluate if arterial inflammation (by PET) correlates with inflammatory cell activation and other measured biomarkers separately. We will then compare the strength of the associations and test their independence. The evaluation of associations will be performed: comparing baseline measurements (SA 2.1), and comparing post-randomization changes (SA2.2).

We expect that LDMTX therapy will improve arterial inflammation and that this mechanistic, proof-of-concept study will demonstrate the importance of inflammation and immune activation in HIV. This would thus form the basis for event-driven trials to evaluate whether anti-inflammatory strategies reduce CVD risk in individuals with treated HIV infection. Accordingly, the study has the potential to shift the paradigm in the approach to treating atherosclerosis in HIV-infected individuals, and potentially in other populations as well.

ELIGIBILITY:
1. Inclusion Criteria:

1.1 HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

NOTE: The term "licensed" refers to a US FDA-approved kit, which is required for all IND studies.

WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

1.2 Currently on continuous ART for ≥24 weeks prior to study entry. This is defined as continuous active therapy for the 24-week period prior to study entry with no treatment interruption longer than 7 consecutive days and a total duration off treatment of no more than 14 days in the 90 days prior to study entry.

1.3 CD4+ T-cell count ≥400 cells/mm3 obtained within 60 days prior to study entry by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.

1.4 HIV-1 RNA level below the limit of quantification using a FDA-approved assay for at least 24 weeks prior to study entry and confirmed within 60 days prior to study entry. The assay used for eligibility can be performed by any US laboratory that has a CLIA certification or its equivalent.

NOTE: Single determinations that are between the assay quantification limit and 200 copies/mL are allowed as long as the preceding and subsequent determinations are below the level of quantification.

1.5 The following laboratory values obtained within 60 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent;

* Fasting glucose <180 mg/dL
* ALT [serum glutamic pyruvic transaminase (SGPT)] <2 times upper limit of normal (ULN)
* AST [serum glutamic oxaloacetic transaminase (SGOT)] <2 x ULN
* Estimated creatinine clearance (CrCl) ≥50 mL/min by Cockcroft-Gault (see section 6.3.5 for CrCl instructions) NOTE: Candidates who are taking TDF as part of their ART regimen must have an estimated CrCl ≥60 mL/min.
* White blood cell (WBC) >3000/mm3
* Hemoglobin >12.0 g/dL
* Platelets >150,000/mm3

1.6 Females subjects who are postmenopausal (i.e., of non-childbearing potential), defined as having either:

1. Appropriate medical documentation of prior hysterectomy and/or complete bilateral oophorectomy (i.e., surgical removal of the ovaries, resulting in "surgical menopause" and occurring at the age at which the procedure was performed), OR
2. Permanent cessation of previously occurring menses as a result of ovarian failure with documentation of hormonal deficiency by a certified healthcare provider (i.e., "spontaneous menopause"). Hormonal deficiency should be properly documented in the case of suspected spontaneous menopause as follows:

   1. If age >54 years and with the absence of normal menses for at least 24 consecutive months: serum follicle stimulating hormone (FSH) level elevated to within the post-menopausal range based on the laboratory reference range where the hormonal assay is performed;
   2. If age ≤ 54 years and with the absence of normal menses for at least 24 consecutive months: Negative serum or urine (β-HCG) performed within 48 hours prior to study entry with concurrently elevated serum FSH level in the post-menopausal range, depressed estradiol (E2) level in the post-menopausal range, and absent serum progesterone level, based on the laboratory reference ranges where the hormonal assays are performed.

1.7 Male subjects must agree not to participate in a conception process (i.e., active attempt to impregnate, sperm donation). If participating in sexual activity that could lead to pregnancy, the male subject must agree to the use of TWO reliable forms of contraceptives simultaneously while on study and for a minimum of 3 months after therapy.

At least TWO of the following contraceptives MUST be used appropriately by male subjects and their female partners:

* Condoms (male or female) with or without a spermicidal agent
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Tubal ligation
* Hormone-based contraceptive

NOTES: Sexual activity that could lead to pregnancy is not applicable to sexual activity with an infertile partner.

Acceptable documentation for the use of two methods of contraceptives is the male subject's report of use of a second form of contraceptive by his female partner.

1.8 Subjects who are not of reproductive potential (defined as women who have been postmenopausal for at least 24 consecutive months or men who have documented vasectomy) are eligible for the study without requiring the use of contraceptives. In order to verify lack of reproductive potential, written documentation or verbal communication by the clinician or clinician's staff of one of the following must be in the source documents:

* Physician report/letter.
* Operative report or other source documentation in the patient record.
* Discharge summary.
* Follicle-stimulating hormone (FSH) measurement elevated into the menopausal range as established by the reporting laboratory.

NOTES: Any statement of self-reported sterility or infertility (or that of a partner's) should be entered into the source document.

Females who report being postmenopausal for at least 24 consecutive months but who do not have documentation of postmenopausal status from a clinician will have the hormonal assessments performed prior to study entry.

1.9 Moderate or high CVD risk defined as:

A) Documented CVD as assessed by meeting at least 1 of 3 criteria below:

1. Coronary artery disease (CAD): prior MI due to atherosclerosis, coronary artery bypass graft surgery, percutaneous coronary intervention, or angiographic CAD with luminal diameter stenosis of at least one coronary artery at least 50%.
2. Cerebrovascular disease: prior ischemic stroke of carotid origin, carotid endarterectomy or stenting, or angiographic carotid stenosis of at least 50%.
3. Peripheral arterial disease: prior lower extremity arterial surgical or percutaneous revascularization procedure, or angiographic lower extremity arterial stenosis of at least 50%.

OR

B) Controlled type II diabetes mellitus (HbA1C ≤8.0% within the past 90 days prior to study entry, regardless of use of medications)

OR

C) Any one of the following CVD risk factors below:

1. Current smoking: subject report of smoking at least a half a pack of cigarettes a day, on average, in the past month.
2. Hypertension (HTN): two consecutive BP readings with either systolic >140 mmHg or diastolic >90 mmHg; or on antihypertensive medications.
3. Dyslipidemia: defined as non-HDL-C >160 mg/dL, regardless of medication use.
4. hsCRP ≥2mg/L

1.10 Men and women age ≥40 years.

1.11 Ability and willingness of subject to provide informed consent.

1.12 For subjects taking tenofovir (TFV) as part of their ART regimen, willingness to conside participate in the PK component of the study.

NOTE: Participation in the PK component is optional but strongly encouraged.

1.13 Completion of the pre-entry FMD assessment.

NOTE: At least one FMD must be performed at the site and confirmed as acceptable by the University of Wisconsin Atherosclerosis Imaging Research Program (UW AIRP) core lab prior to study entry.

1.14 Additional Inclusion criteria for the Imaging sub-study:

To be eligible for the PET/CT Imaging sub-study, the subject must:

A) Be a participant in the Parent Study B) Not yet have received study drug C) Be able to undergo imaging prior to randomization

2. Exclusion Criteria:

2.1 Acute or serious illness requiring systemic treatment and/or hospitalization within 60 days prior to study entry.

NOTE: Treatment must have ended at least 60 days prior to study entry for eligibility.

2.2 Documentation of any CDC category C AIDS-indicator condition [78] or oropharyngeal candidiasis (thrush) within 90 days prior to study entry.

2.3 Receipt of antibiotic therapy within 30 days prior to study entry.

2.4 Latent TB infection (defined as a positive PPD ≥5 mm, positive interferon-gamma release assay, or positive T-spot test at any time in the past) or evidence of latent TB on the screening chest x-ray that has not been completely treated or was treated within the past 6 months prior to study entry .

2.5 TB disease requiring treatment within 48 weeks prior to study entry.

2.6 Life-threatening fungal infection requiring treatment, in the opinion of the site investigator, within 48 weeks prior to study entry.

2.7 Herpes-zoster viral infection requiring treatment within 90 days prior to study entry.

2.8 A history of or current, active hepatitis B infection defined as positive hepatitis B surface antigen test or positive HBV DNA in subjects with isolated HBcAb positivity, defined as negative HBsAg, negative HBsAb, and positive HBcAb within 24 weeks prior to study entry.

NOTE: Subjects who are positive for hepatitis B surface antigen but who are HBV DNA negative are permitted in the study.

2.9 Chronic hepatitis C infection defined as a positive hepatitis C antibody and positive hepatitis C RNA at any time prior to study entry.

NOTE: Subjects who are positive for hepatitis C antibody but who are HCV RNA negative are permitted in the study.

2.10 Previously diagnosed myelodysplasia syndrome.

2.11 Treated lymphoproliferative disease ≤5 years prior to study entry.

2.12 Clinically significant lung disease on the screening chest x-ray that, in the opinion of the site investigator, places the subject at increased risk of lung toxicity (e.g., history of pulmonary fibrosis, interstitial lung disease, or pulmonary lymphoproliferative disease).

2.13 Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry.

2.14 Change in the ART regimen in the 12 weeks prior to study entry or intended modification of ART during the study.

NOTE: Modifications of ART doses during the 12 weeks prior to study entry are permitted. In addition, the change in formulation (e.g., from standard formulation to fixed-dose combination) is allowed within 12 weeks prior to study entry. A within class single drug substitution (e.g., switch from nevirapine to efavirenz or from atazanavir to darunavir) is allowed within 12 weeks prior to study entry, with the exception of a switch from any other NRTI to abacavir. No other changes in ART in the 12 weeks prior to study entry are permitted.

2.15 Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.

2.16 Average daily consumption of three or more alcoholic beverages for 4 weeks prior to study entry or intention to consume an average of two or more alcoholic beverages a day during the study.

NOTE: An alcohol-containing beverage is defined as 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits.

2.17 Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

2.18 Changes in lipid-lowering or antihypertensive medication within 90 days prior to study entry or expected need to modify these medications during the study.

NOTE: Lipid-lowering medication includes: statins, fibrates, niacin (dose ≥250 mg daily), and fish-oil/omega 3 fatty acids (dose >1000 mg of marine oils daily).

2.19 Vaccination (e.g., influenza, pneumococcal polysaccharide) within 14 days prior to study entry.

2.20 Anticipated need to receive vaccination (e.g., influenza, pneumococcal polysaccharide) within 1 week prior to week 4, 12, 24, or 36 study visits.

2.21 Excess extracompartmental fluids including ascites, pericardial fluid, and pleural effusions which, in the opinion of the study investigators, would result in difficulty in monitoring the dose of MTX.

2.22 Use of drugs that alter folic acid metabolism such as trimethoprim/sulfamethoxazole or reduce tubular excretion such as probenecid within 14 days prior to study entry.

2.23 New York Heart Association Class IV congestive heart failure.

2.24 Diabetes mellitus with HbA1C >8.0% within the past 90 days prior to study entry.

2.25 Patients who report any significant radiation exposure over the course of the year prior to randomization. Significant exposure is defined as:

i) More than 2 PCI within 12 months of randomization ii) More than 2 myocardial perfusion studies within the past 12 months iii) More than 2 CT angiograms within the past 12 months iv) Any subjects with history of radiation therapy.

2.26 Current daily use of insulin.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subset of individuals enrolled in A5314 who undergo PET/CT imaging.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Tawakol, MD, Principal Investigator — Massachusetts General Hospital and Harvard Medical School
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Methotrexate | Placebo
Started | 13 | 22
Completed | 12 | 16
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — could not schedule imaging in time | 0 | 2
Not completed — Other | 0 | 1
Not completed — Not randomized. Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Methotrexate | Placebo | Total
Number analyzed (Participants) | 12 | 16 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [51 to 59.5] | 55.5 [50.5 to 63.5] | 54.5 [50.5 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 12 | 13 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial FDG Uptake (From Baseline) in the Most Diseased Segment
Description: Arterial FDG Uptake provides a measure of inflammation in the artery wall.
  TBR is target-to-background ratio (a measure of the ratio of the activity in the vessel wall divided by the blood background). A negative number for the change in TBR implies a reduction in activity over time.
  The most diseased segment is the approx 1-cm section of the vessel with the highest activity at baseline.
  The results are expressed as the change in the median value, of the TBR, from baseline to week 24
Time Frame: baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: TBR
Arm/Group | Low Dose Methotrexate | Placebo
Number analyzed (Participants) | 12 | 16
TBR | -0.126 [-0.41 to 0.258] | 0.026 [-0.176 to 0.438]

2. Secondary Outcome: Change in Arterial FDG Uptake (From Baseline) in the Aorta
Description: Arterial FDG Uptake provides a measure of inflammation in the artery wall.
  TBR is target-to-background ratio (a measure of the ratio of the activity in the vessel wall divided by the blood background). A negative number for the change in TBR implies a reduction in activity over time.
  The entire ascending aorta is used for this analysis.
  The results are expressed as the change in the median value, of the TBR, from baseline to week 24
Time Frame: baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: TBR
Arm/Group | Low Dose Methotrexate | Placebo
Number analyzed (Participants) | 12 | 16
TBR | -0.064 [-0.327 to 0.113] | 0.063 [-0.13 to 0.425]

ADVERSE EVENTS:
Arm/Group | Low Dose Methotrexate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 0/12 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes